CLINICAL TRIAL: NCT03917108
Title: Assessment of Technique Sensitivity and Gingival Health in Management of Cervical Lesions Performed Using Subgingival Clamp Versus Retraction Cord: A Randomized Controlled Clinical Trial
Brief Title: Subgingival Clamp Versus Retraction Cord in Cervical Lesions in Term of Technique Sensitivity and Gingival Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Hamada Ahmed Shehab Eldin, principal investigator in Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 603
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Gingival Retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- retraction cord (Active Comparator)
  Interventions: Device: retraction cord
- subgingival clamp (Other)
  Interventions: Device: subgingival clamp

INTERVENTIONS:
Device: retraction cord — retraction cord ( Ultra dent sizes #0, #00, #000 ) is placed in the gingival sulcus using blunt instrument and using cotton roll isolation.
  Arms: retraction cord
Device: subgingival clamp — subgingival clamp (KSK clamps W8A, #44, #42, #43) or (Brinker clamps B5, B6) is placed to retract the gingiva with rubber dam isolation
  Arms: subgingival clamp

SUMMARY:
assessing subgingival clamp in handling and retracting the gingival tissue at the cervical area to see its effect on the gingival health and its technique sensitivity compared to the most commonly used method (retraction cord), as gingival displacement for cervical restorations affects smile and therefore patient satisfaction with the result.

DETAILED DESCRIPTION:
Gingival displacement for restoring cervical lesions using retraction cord or subgingival clamp with their technique sensitivity affects the smile as they may cause gingival bleeding, laceration or recession and therefore affects patient satisfaction. There are several methods to achieve retraction; retraction cord is the most commonly used method. It controls the soft tissue displacement, gingival bleeding and expose the margins which provide good visualization and access.

They are effective and safe if the gingiva is healthy, also inexpensive retraction method. However, the use of retraction cord has some disadvantages like: it is time consuming, may cause gingival recession after healing and bleeding after removal, its application needs practice and skill as improper handling of the cord can cause traumatic injuries, gingival recession and marginal exposure of the restoration, it may cause postoperative discomfort and pain for the patient and finally leaving the retraction cord for long time or forgetting to remove it from the sulcus can cause permanent damage to the gingival tissue.

Using gingival retracting clamps with rubber dam isolation prevent the gap caused around the teeth due to vertical and horizontal tissue displacement occurred beneath the area of dento-gingival attachment upon the application of the retraction cord. Also, after clamp stabilization in position, it prevents accidental slippage and trauma to surrounding soft tissue during the restorative procedure. They also provide maximum tissue retraction without laceration of gingival tissues. Also, their availability in different sizes and shapes provide a good adaptation to any tooth configuration and any inaccessible area.

ELIGIBILITY:
Inclusion Criteria:

* Subject not less than 18 years of age.
* Males or females.
* Have at least one carious or non-carious cervical lesion.
* Cervical lesions should be equi-gingival or subgingival.
* Can comply to oral hygiene measures or with good oral hygiene.
* Have sufficient cognitive ability to understand consent procedures.
* Vital upper or lower teeth with no signs or symptoms of irreversible pulpitis.
* Clinically healthy gingiva and periodontium.
* No evidence of attachment loss, bleeding on probing, or plaque accumulation.

Exclusion criteria:

* Exclusion Criteria:
* Patients less than 18 years old.
* Disabilities (mental health conditions, intellectual disability and physical disabilities).
* Systemic diseases or severe medically compromised. (Cardiovascular disorder, diabetes, -hypertensive, epileptic.
* Lack of compliance.
* Gingival hyperplasia, blood disorder.
* Attachment loss signs of periodontal disease.
* Patients contra-indicated for rubber dam placement (Asthmatic patient, mouth breather, -- partially erupted tooth, extremely malposed teeth and latex allergy).
* Periapical pathosis or signs of pulpal posterior or anterior pathology.
* Non-vital tooth.
* Endodontically treated tooth.
* Sever periodontal affection.
* Tooth indicated for extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Time of application | Immediately after application
  Assessed using timer and the measuring unite is seconds
Number of patients need local anesthesia | Immediately after application
  It will be measured by patient self assessment for the need of local anesthesia through a Yes/No question
Degree of isolation from cervical fluids | Immediately after application
  Presence of cervical fluids will be assessed visually using magnifying loup with a Yes/No result
Degree of patient satisfaction | Immediately after application
  Using visual analogue scale (units on scale from 0-10)

SECONDARY OUTCOMES:
Pink esthetics evaluation | 4 month
  Using a pink esthetic score with a grades from 0-2
Amount of gingival bleeding | 4 month
  Assessed using a score for gingival hemorrhage from 0 -2
Presence of gingival laceration | 4 month
  Occurence of gingival laceration assessed visually using magnifying loup with a Yes/No result
Degree of gingival sensitivity | 4 month
  Assessed using visual analogue scale (units on scale from 0-10)